CLINICAL TRIAL: NCT02015013
Title: Hematopoietic Stem Cell Mobilization in Idiopathic CD4 Lymphocytopenia Patients and Healthy Controls for the Study of T Cell Maturation and Trafficking in Murine Models
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 140020; 14-I-0020
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-11-24

CONDITIONS: Idiopathic CD4-Positive; T-Lymphocytopenia
Keywords: Leukapheresis; Progenitor Cells
MeSH Terms: conditions — T-Lymphocytopenia | interventions — Filgrastim; plerixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Filgrastim (Experimental): ICL and healthy volunteers will be given 10 microgram/kg daily for 5 days administered according to a vial-based algorithm to reduce wastage and increase the G-CSF dose given to lighter-weight donors to improve CD34+ yields
  Interventions: Biological: Filgrastim
- Plerixafor (Experimental): ICL and healthy volunteers will be given 0.24 mg/kg as a single dose (maximum dose: 40 mg) 11 hours prior to apheresis
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Biological: Filgrastim — 10 microgram/kg daily for 5 days, Subcutaneous injection.
  Arms: Filgrastim
Drug: Plerixafor — IV injection 0.24 mg/kg as a single dose, 11 hours prior to apheresis
  Arms: Plerixafor

SUMMARY:
Idiopathic CD4 lymphocytopenia (ICL) is a rare syndrome defined by consistently low CD4 T cell counts (<300/mm3) without evidence of HIV infection or other known immunodeficiency. Patients with ICL are at risk for opportunistic infections typically associated with HIV/AIDS such as disseminated cryptococcal infection and severe human papillomavirus-related dysplasia. More than 20 years since the description of ICL, its etiology, pathogenesis, and management remain unclear. In this study we propose to administer the combination of granulocyte colony stimulating factor (G-CSF) and plerixafor to ICL patients and healthy volunteers with the objective of harvesting mobilized CD34+ hematopoietic progenitor cells (HPCs) by apheresis for transfer into immunocompromised mice and for study with in vitro assays. The mice studies would serve to investigate thymic development, survival, and trafficking of the mobilized human cells within murine lymphoid and non-lymphoid organs.

HPCs are used for various therapies and there is an increasing use of agents that stimulate the bone marrow to produce progenitor cells and move them into the bloodstream where they may be harvested by apheresis. Not all patients respond to GCSF with vigorous HPC mobilization. The binding of chemokine receptor CXCR4 to stromal cell derived factor (SDF-1 or CXCL12) is an important interaction between a hematopoietic progenitor cell and its marrow environment. Plerixafor is a CXCR4 inhibitor which blocks binding to SDF-1 resulting in the release of hematopoietic progenitor cells (CD34+) into peripheral circulation. In pharmacodynamic studies of plerixafor in conjunction with G-CSF compared to G-CSF and placebo, a two-fold increase in CD34+ cell count was observed.

Due to the important role CXCR4 plays in immune cell trafficking and its potential role in the pathogenesis of ICL, we propose as a secondary objective to assess peripheral CD4 T cell and CD34+ hematopoietic progenitor cell numbers and functions in ICL patients compared to controls following G-CSF and plerixafor administration.

Study participants will be screened within 12 weeks prior to the study period. Eligible participants will receive G-CSF for 5 days with hospitalization on Day 4 for plerixafor injection followed by apheresis on Day 5. Participants will return for examinations and blood draws on Days 8 and 12.

DETAILED DESCRIPTION:
Idiopathic CD4 lymphocytopenia (ICL) is a rare syndrome defined by consistently low CD4 T cell counts (<300/3microL) without evidence of HIV infection or other known immunodeficiency. Patients with ICL are at risk for opportunistic infections typically associated with HIV/AIDS such as disseminated cryptococcal infection and severe human papillomavirus-related dysplasia. More than 20 years since the description of ICL, its etiology, pathogenesis, and management remain unclear. In this study we propose to administer the combination of granulocyte colony stimulating factor (G-CSF) and plerixafor to ICL patients and healthy volunteers with the objective of harvesting mobilized CD34+ hematopoietic progenitor cells (HPCs) by apheresis for transfer into immunocompromised mice and for study with in vitro assays. The mice studies would serve to investigate thymic development, survival, and trafficking of the mobilized human cells within murine lymphoid and non-lymphoid organs.

HPCs are used for various therapies and there is an increasing use of agents that stimulate the bone marrow to produce progenitor cells and move them into the bloodstream where they may be harvested by apheresis. Not all patients respond to GCSF with vigorous HPC mobilization. The binding of chemokine receptor CXCR4 to stromal cell derived factor (SDF-1 or CXCL12) is an important interaction between a hematopoietic progenitor cell and its marrow environment. Plerixafor is a CXCR4 inhibitor which blocks binding to SDF-1 , resulting in the release of HPCs (CD34+) into peripheral circulation. In pharmacodynamic studies of plerixafor in conjunction with G-CSF compared to G-CSF and placebo, a two-fold increase in CD34+ cell count was observed.

Due to the important role CXCR4 plays in immune cell trafficking and its potential role in the pathogenesis of ICL, we propose as a secondary objective to assess peripheral CD4 T cell and CD34+ hematopoietic progenitor cell numbers and functions in ICL patients compared to controls following G-CSF and plerixafor administration.

Study participants will be screened within 12 weeks prior to the study period. Eligible participants will receive G-CSF for 5 days with hospitalization on Day 4 for plerixafor injection followed by apheresis or large volume blood draw (120 cc) on Day 5. Participants will return for examinations and blood draws on Days 8 and 12.

ELIGIBILITY:
* INCLUSION CRITERIA

ICL patients:

1. Documented history of idiopathic CD4 lymphocytopenia as defined by CD4 T cell count <300 cells/microL or <20% of total T lymphocytes on 2 occasions at least 6 weeks apart in the absence of any illness or medications accounting for CD4 lymphocytopenia. Although the protocol will primarily enroll ICL patients who are lymphopenic at the time of enrollment, up to three patients who had clear documentation of ICL in the past and are currently not lymphopenic may still be enrolled for comparative purposes.
2. Hemoglobin greater than or equal to 9 g/dL
3. Human T-lymphotropic virus Type 1 (HTLV-1) and HTLV-2 seronegative
4. Persons with documented history of ICL in whom genetic analysis revealed inherited defects that are either known or suspected to be involved in development, maturation, or homeostasis of hematopoietic cells.

Healthy volunteers: white blood cell count >2500/microL and hemoglobin greater than or equal to 12.5 g/dL

ICL patients and healthy volunteers:

1. Age 18-65 years
2. Weight at least 50 kg but less than 167 kg and <175% ideal body weight (due to lack of data regarding appropriate dosing of plerixafor)
3. Ability to give informed consent
4. Capacity and willingness to adhere to study procedures, including scheduled follow-up visits
5. Willingness to have blood samples stored for future research
6. Willingness to undergo HLA testing
7. Willingness to be hospitalized for approximately 24 hours
8. Established primary care provider
9. HIV-1 and HIV-2 seronegativity and plasma HIV-1 RNA polymerase chain reaction (PCR) below the limit of detection
10. Adequate venous access to allow leukapheresis without use of a central line or a large volume blood draw
11. Participant agrees to be heterosexually inactive or consistently use effective birth control (e.g., barrier methods, oral contraceptives, intrauterine devices, vasesctomy) for the duration of study participation and for approximately 8 weeks after the last dose of G-CSF. This is necessary for both male and female participants.
12. For women of childbearing potential:

    1. Negative serum or urine pregnancy test

EXCLUSION CRITERIA

1. Active uncontrolled infection at the time of enrollment
2. Current autoimmune conditions requiring systemic (oral, injection, or other parenteral) therapy
3. History of vasculitis
4. Current or history of hematologic or lymphoid malignancy (leukemia)
5. History of splenomegaly or current splenomegaly on exam or ultrasound (for ICL patients)
6. History of hypersensitivity to plerixafor and/or G-CSF
7. Systemic immune-modulatory agent within the past 6 months
8. Thrombocytopenia (platelets <100,000 cells/microL)
9. Hepatitis B and C seropositivity (HBsAg positive and anti-HCV positive) Need for anticoagulant medication (e.g., warfarin, heparin), other than aspirin, clopidogrel, or other antiplatelet agent
10. Creatinine clearance <50 mL/min including end-stage renal disease requiring hemodialysis
11. Symptomatic coronary artery disease
12. Uncontrolled hypertension (i.e., resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >90 mmHg) despite pharmacologic antihypertensive treatment confirmed with a second blood pressure measurement done later on the same day
13. Cardiac, pulmonary, thyroid, renal, hepatic, neurological (central or peripheral) disease or disorder of hemostasis requiring therapy and considered to be significant by the protocol team
14. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
15. Currently receiving lithium due to contraindication of co-administration of G-CSF with lithium
16. Past or current psychiatric illness that, in the opinion of the investigator, would interfere with protocol adherence or the ability to give written informed consent
17. Any illness or condition that, in the opinion of the investigator, may substantially increase the risk associated with participation in the study or compromise the scientific objectives
18. Participation in a clinical protocol which includes an intervention that, in the opinion of the investigator, may affect the results of the current study
19. Previous history of anaphylactic reaction to aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
20. Female of child-bearing potential who is breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
To mobilize CD34+ HPCs in ICL patients and healthy volunteers for collection and transfer into immunocompromised mice to investigate thymic development, survival, and trafficking of these cells in murine lymphoid and non-lymphoid organs | Throughout the study
  Collection of CD34+ cells from ICL patients and healthy volunteers to investigate thymic development, survival, and trafficking of these mobilized cells in the lymphoid and non lymphoid organs of mice.

SECONDARY OUTCOMES:
To assess peripheral CD4 T cell and CD34+ HPC numbers and functions in ICL subjects compared to controls following G CSF and plerixafor administration | Throughout the study
  Collection of peripheral CD4 T cells and CD34+ HSCs for comparison of number and function of these cell types in ICL patients and healthy volunteers. The function of progenitor cells will be measured as multipotency.

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Anyone who wishes to access the data on clinical trials website

REFERENCES:
- [Background] Isgro A, Sirianni MC, Gramiccioni C, Mezzaroma I, Fantauzzi A, Aiuti F. Idiopathic CD4+ lymphocytopenia may be due to decreased bone marrow clonogenic capability. Int Arch Allergy Immunol. 2005 Apr;136(4):379-84. doi: 10.1159/000084258. Epub 2005 Mar 2. PMID 15746558
- [Background] Fruhwirth M, Clodi K, Heitger A, Neu N. Lymphocyte diversity in a 9-year-old boy with idiopathic CD4+ T cell lymphocytopenia. Int Arch Allergy Immunol. 2001 May;125(1):80-5. doi: 10.1159/000053800. PMID 11385292
- [Background] Hubert P, Bergeron F, Ferreira V, Seligmann M, Oksenhendler E, Debre P, Autran B. Defective p56Lck activity in T cells from an adult patient with idiopathic CD4+ lymphocytopenia. Int Immunol. 2000 Apr;12(4):449-57. doi: 10.1093/intimm/12.4.449. PMID 10744646
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-I-0020.html